CLINICAL TRIAL: NCT03204539
Title: INdividualized ITI Based on Fviii(ATE) Protection by VWF (INITIATE)
Brief Title: INdividualized ITI Based on Fviii(ATE) Protection by VWF
Acronym: INITIATE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Termination of funding from sponsor.
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 988465
Record Dates: First submitted 2017-06-13; First posted 2017-07-02 (Actual); Results first posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Hemophilia A With Inhibitor; Hemophilia A
Keywords: inhibitor; Factor VIII inhibitor
MeSH Terms: conditions — Hemophilia A | interventions — von Willebrand Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alternative Treatment (Experimental): Half of the participants will be randomized to blinded individualized lot selection for ITI.
  Interventions: Drug: Wilate
- Standard Treatment (Other): The other half of the participants will receive random lot selection for ITI.
  Interventions: Drug: Wilate

INTERVENTIONS:
Drug: Wilate — Wilate® is a high-purity (i.e. 100 IU FVIII/mg total protein) pdVWF/FVIII complex concentrate.Wilate® possesses all the important features asked for in ITI, namely high purity, a very high pathogen safety profile, and an excellent protection of its FVIII by VWF - all achieved through unique, novel, and innovative techniques.

SUMMARY:
The primary goal of the INITIATE trial is to compare the clinical outcome of individualized lot selection to random lot selection utilizing one plasma-derived von Willebrand factor (VWF)/coagulation factor (FVIII) complex concentrate for immune tolerance induction (ITI) in subjects with congenital Hemophilia A, FVIII activity ≤2%, and a historical high-titer inhibitor [≥5 Bethesda Unit (BU)].

DETAILED DESCRIPTION:
Participants will be randomized on a one-to-one basis between one of two study arms, individualized lot selection (alternative treatment arm) and random lot selection (standard treatment arm, current US clinical practice in ITI). Study sites, participants, and investigators will be blinded to the treatment status assigned.

Alternative treatment arm:

Half of the participants will be randomized to blinded individualized lot selection for ITI. The target initial dose of FVIII for ITI is ~200 IU/kg/day intravenously. The suggested maximum dose is 20,000 IU/day. Investigators may adjust the dose to a minimum dose of 150 units/kg if infusion volume is not feasible in patients without central venous access or in patients with von Willebrand factor levels >250%. Splitting dose into two infusions per day must be approved by the Steering Committee, and if approved, will be considered a protocol deviation. Wilate® will be the VWF/FVIII complex concentrate (Octapharma USA, Inc., U.S. License No. 1646) prescribed for ITI.

Individualized lot selection will be performed according to a modified Oxford method in a central laboratory, by testing subject's plasma against 4-6 lots of Wilate® and selecting the one with the highest residual FVIII (lowest Oxford titer) activity remaining after incubation. The same lot will be used throughout the entire ITI course for each subject. If the selected lot is depleted prior to the completion of ITI, a second individualized lot selection will be performed using the original plasma sample provided at baseline.

Each Wilate® batch includes 1.6-1.8 million IU and is expected to last for about 3-57 months depending on the weight of the subject and prescribed dose.

Standard treatment arm:

The other half of the participants will receive random lot selection for ITI. The dose and concentrate used will be the same. Concentrate will be randomly selected from available Wilate® lots. The same lot will be used throughout the entire ITI course for each subject. If the random lot is depleted prior to the completion of ITI, a second lot will be randomly selected. In both cases the random lot will be tested against subject's plasma to measure the residual FVIII activity left after incubation but this result will not affect lot selection.

The primary hypothesis is that the time to negative inhibitor (<0.6 BU) will be shorter with individualized lot selection compared to random lot selection and that this will impact monthly break-through bleeding and reduce costs.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of congenital Hemophilia A and baseline FVIII ≤2%.
2. Weight ≥ 5 kg
3. History of FVIII inhibitor titer ≥5 BU
4. Current FVIII inhibitor titer ≥5 BU or ≥0.6 BU and failed ITI defined by FVIII recovery <66% normal and half-life <6 hours
5. Adequate venous access for daily concentrate infusions
6. For participants <18 years, a parent or guardian willing and able to provide informed consent with verbal or written assent from the child if require by the local institution. For participants ≥18 years, a willingness and ability to provide informed consent from the subject.
7. Ability to comply with study related treatments, evaluations, and follow-up.

Exclusion Criteria:

1. Acquired hemophilia
2. Congenital or acquired bleeding disorder in addition to Hemophilia A
3. ITI factor replacement regimen within the past one month unless there is clear evidence of ITI failure with no reduction in inhibitor titer over the past two months
4. HIV positive with viral load ≥200 particles/μL or ≥400,000 copies/mL
5. Rituximab within the past 3 months
6. IVIG within the past 1 month
7. Treatment with other immunosuppressive drugs within the past 1 month (excluding intermittent steroid use for asthma)
8. Concomitant experimental treatment
9. History of hypersensitivity to plasma-derived VWF- or FVIII-containing concentrates
10. Elective surgery planned in the next 6 months (excluding vascular access procedure)
11. Any condition or chronic illness, which in the opinion of the investigator makes participation ill-advised
12. Inability or unwillingness to complete required screening, follow-up, and exit studies

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 1 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California, Davis, Sacramento, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Tulane University, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only 1 participant enrolled, but did not complete study due to early study termination.
Period: Overall Study
Arm/Group | Alternative Treatment | Standard Treatment
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Loss of funding | 0 | 1

BASELINE CHARACTERISTICS:
Population: Only 1 participant enrolled (standard treatment arm), and did not complete study due to loss of funding.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alternative Treatment | Standard Treatment | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Customized [Number; unit: years]
  Age |  | 5 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 1 | 1
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 1 | 1
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Negative Inhibitor
Description: This endpoint was chosen because a shorter time to negative inhibitor should decrease monthly break-through bleeding frequency in the early phase of ITI
Time Frame: completion of immune tolerance induction, up to 18 months
Population: Study terminated, and no participants completed study. No outcome measure data to report.
Arm/Group | Alternative Treatment | Standard Treatment
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time to Achieve Partial and Complete Success
Description: Secondary endpoints include time to achieve partial and complete success as defined according to the following criteria:
  * Inhibitor titer <0.6 BU.
  * Incremental in vivo FVIII recovery in the normal range [≥66% of normal (1.5% per IU/kg), equal to 0.99%per IU/kg] with samples taken prior to and 15 or 30 minutes after concentrate treatment. The recovery assessment should be done without any wash-out period.
  * Half-life of FVIII >6 hours. The half-life assessment should be done in a non-bleeding status without any wash-out period.
  Complete Success (CS) of ITI:
  All three criteria above met.
  Partial Success (PS) of ITI:
  The first two of the three criteria above met.
  Partial Response (PR) of ITI:
  One of the three criteria above met.
  Partial Failure (PF) of ITI:
  Inhibitor still present, but titer is decreased to <5 BU in contrast to ≥5 BU before start.
  Complete Failure (CF) of ITI:
  None of the above mentioned criteria met, and the inhibitor titer is still ≥5 BU.
Time Frame: completion of immune tolerance induction, up to 18 months
Population: Study terminated, and no participants completed study. No outcome measure data to report.
Arm/Group | Alternative Treatment | Standard Treatment
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Absence of Relapse, up to 12 Months After Achievement of Complete or Partial ITI Success
Time Frame: one year after completion of immune tolerance induction, up to 30 months
Population: Study terminated, and no participants completed study. No outcome measure data to report.
Arm/Group | Alternative Treatment | Standard Treatment
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: The Number of Break-through Bleeding Events During the Course of ITI-treatment·
Time Frame: completion of immune tolerance induction, up to 18 months
Population: Study terminated, and no participants completed study. No outcome measure data to report.
Arm/Group | Alternative Treatment | Standard Treatment
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Cost of ITI - Including Bleeding Control Using Bypassing Agents Prior to Start and During ITI
Time Frame: completion of immune tolerance induction, up to 18 months
Population: Study terminated, and no participants completed study. No outcome measure data to report.
Arm/Group | Alternative Treatment | Standard Treatment
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Subject Quality of Life
Description: measured with the Haemo-QOL questionnaire
Time Frame: completion of immune tolerance induction, up to 18 months
Population: Study terminated, and no participants completed study. No outcome measure data to report.
Arm/Group | Alternative Treatment | Standard Treatment
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Subject Compliance With ITI Treatment Regimen
Description: We will be looking at drug accountability reports/ logs which will reflect each subject's usage of Wilate
Time Frame: completion of immune tolerance induction, up to 18 months
Population: Study terminated, and no participants completed study. No outcome measure data to report.
Arm/Group | Alternative Treatment | Standard Treatment
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: The Impact of Inhibitor Titer at Start of ITI and During the Course of ITI, Including the Peak Titer of the Inhibitor
Time Frame: completion of immune tolerance induction, up to 18 months
Population: Study terminated, and no participants completed study. No outcome measure data to report.
Arm/Group | Alternative Treatment | Standard Treatment
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Understand Other Factors Related to ITI Success Using Additional Biologic Assays
Description: If subject consents, the following assays will be performed:
  epitope mapping immunogenotyping/HLA genotyping FVIII genetic testing
Time Frame: screening/baseline
Population: Study terminated, and no participants completed study. No outcome measure data to report.
Arm/Group | Alternative Treatment | Standard Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Only 1 participant enrolled in study (Standard treatment arm) due to loss of funding.
Arm/Group | Alternative Treatment | Standard Treatment
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/1
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alternative Treatment (N=0) | Standard Treatment (N=1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alternative Treatment (N=0) | Standard Treatment (N=1)
Fever (Infections and infestations) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/39/NCT03204539/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT03204539/ICF_001.pdf